## Statistical Analysis Plan

Grant Title: Peer Based Suicide Prevention

ClinicalTrials.gov ID: NCT04222673

Sponsor: VA Office of Research and Development

Document date: March 8, 2022

Given the small sample size and recommendations for pilot studies,  $^{36}$  quantitative analyses were descriptive (e.g., frequencies, means) and based on the Reliable Change Index (RCI) $^{37}$  for each participant for each outcome measure. The RCI is used to determine whether pre- to post-score differences are statistically reliable and to categorize changes as either improved, deteriorated, or indeterminate.  $^{38}$  A statistical threshold of RCI score  $z = \pm 1.96$  and p < .05 was used to establish clinical significance.